CLINICAL TRIAL: NCT02683915
Title: Acute Kidney Injury in Asphyxiated Infants Treated by Therapeutic Hypothermia
Brief Title: Reno-protective Effect of Brain Cooling in Newborn With Hypoxia
Status: Completed | Type: Observational
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Assistant Professor of pediatrics, Mansoura University Children Hospital
Other Study IDs: MS-602
Record Dates: First submitted 2016-02-03; First posted 2016-02-17 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Acute kidney injury; Perinatal asphyxia; Therapeutic hypothermia; Serum NGAL; Serum cystatin-C
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Acute Kidney Injury | interventions — Hypothermia, Induced; Cool-Down Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Therapeutic hypothermia: Infants in cooled group will be fitted a cooling cap (Olympic Medical Cool Care System, Olympic Medical) around the head for 72 h. infants will be nursed under a radiant overhead heater, which is servo-controlled to the infant's abdominal skin temperature and adjusted to maintain the rectal temperature at 33.5-34.5ºC. At the end of the 72 h cooling period, the infants will be slowly rewarmed at no more than 0•5ºC /h until their temperature become within normal temperature range (36.5-37.5ºC).
  Interventions: Procedure: Therapeutic hypothermia
- Non-cooled group: Infants in the non-cooled group received the current standard of care and will be placed under radiant heaters or in incubators, which are servo-controlled according to the abdominal skin temperature to maintain the rectal temperature at 37.0± 0.2°C.

INTERVENTIONS:
Procedure: Therapeutic hypothermia — Infants in cooled group will be fitted a cooling cap (Olympic Medical Cool Care System, Olympic Medical) around the head for 72 h. infants will be nursed under a radiant overhead heater, which is servo-controlled to the infant's abdominal skin temperature and adjusted to maintain the rectal temperature at 33.5-34.5ºC. At the end of the 72 h cooling period, the infants will be slowly rewarmed at no more than 0•5ºC /h until their temperature become within normal temperature range (36.5-37.5ºC).
  Other Names: Cooling
  Groups: Therapeutic hypothermia

SUMMARY:
This study aims to determine the effect of therapeutic hypothermia on reducing AKI in term and late-preterm infants with hypoxic ischemic encephalopathy as estimated by measurment of serum(s) neutrophil gelatinase-associated lipocalin(NGAL) and serum (s) cystatin-C.

DETAILED DESCRIPTION:
The study will be conducted at the NICU of Mansoura University children's Hospital and regional General Hospital where brain cooling is not available.

Infants will be identified in the delivery room or the NICU based on a per-specified inclusion and exclusion criteria. The admitting physician will inform the study team upon admitting the infants to prepare for obtaining consent form.

When a patient is admitted and satisfies the inclusion criteria, one of the investigators or delegate will approach the parent(s). Patient identification will be done by admitting residents or the nurse practitioners. Parents will be approached by the residents or the nurse practitioners while the signature of the consent form in case of agreement will be obtained by one of the investigators who are not responsible about the care of the infant. Using language understandable to the parent(s), the study protocol will be described in detail outlining the procedure and describing any potential risks. All parents will be specifically informed that a decision not to participate in the research study will in no way compromise their child's care. If the parent(s) agree that their child participate in the study, written informed consent will be obtained. A copy of the consent form will be kept with the investigators.

Infants will be classified into two groups, either group 1 (Cooled group) or group 2 (Non-cooled group) who missed opportunity to be identified within proper time.Categorization will be center-based according to the feasibility of cooling devices at proper time (the first 12 hours of the baby's life).

Group 1 (Cooled group) Cooling procedure We will fit a cooling cap (Olympic Medical Cool Care System, Olympic Medical) around the head for 72 h. The system consists of a small thermostatically controlled cooling unit with a pump that circulated water through the cap. The initial water temperature is set between 8°C and 12°C. All infants will be nursed under a radiant overhead heater, which is servo-controlled to the infant's abdominal skin temperature and adjusted to maintain the rectal temperature at 33.5-34.5ºC. Adjustments will be made to the cooling cap water temperature to stay within these limits. At the start of hypothermia, the overhead heater will be turned off for 20-30 min to accelerate cooling, and then turned back on once the rectal temperature had fallen to 35.5ºC.

Rewarming procedure At the end of the 72 h cooling period, the infants will slowly rewarmed at no more than 0.5ºC /h until their temperature was within normal temperature range (36.5-37.5ºC). The overhead heater can be adjusted as needed, to rewarm the infant. The infant's temperature will be be carefully monitored for at least 4 hours to prevent rebound hyperthermia, as this might be detrimental.

Group 2 (Non-cooled group):

Infants in the non-cooled group received the standard of care and will placed under radiant heaters or in incubators, which will be servo-controlled according to the abdominal skin temperature to maintain the rectal temperature at 37.0± 0.2°C.

Laboratory test results Serum creatinine, electrolyte levels, and liver function tests will be assessed before the start of cooling (baseline); at 72 during cooling; and then on days and 10 of life as clinically indicated. Blood sample for sNGAL and cystatine C will be obtained at Day 1, 4 and 10 of life.

Statistical Analysis Statistical analysis will be performed using SPSS statistical software (version 16; SPSS, Chicago, Illinois). Student-t test or Mann-Whitney test will be used to compare continuous variables and Chi-square test or Fisher's exact test will be used for categorical variables. The diagnostic accuracy of the sNGAL and cystatine C tested in this study for identifying AKI will be evaluated by constructing receiver operating characteristics (ROC) curves. A p-value of <0.05 is considered to be statistically significant. All data will be expressed as mean ± standard deviation unless otherwise stated.

ELIGIBILITY:
Inclusion criteria:

1. Full term newborn exposed to peri-natal asphyxia
2. Presented by signs of hypoxic ischemic encephalopathy (Sarnat grade II or III)

Exclusion criteria:

1. Major intracranial haemorrhage
2. Birth weight less than 1800 g.
3. Major congenital anomalies including:

   1. Chromosomal anomalies.
   2. Congenital heart disease.
   3. Congenital diaphragmatic hernia.
   4. Congenital hydrocephalus and neural tube defects.
   5. Intestinal atresia, tracheooesophageal fistulas, and omphalocele.

Ages: 30 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants will be enrolled into two groups either group 1(cooled group) if identified within 12 hours of age and admitted at hospital with a validated cooling facility or group 2(non cooled group) if identified older than 12 hours of age or admitted at hospital out of reach of a validated cooling facility (cooling still not governmentally submitted in Egypt at wide scale).
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 15 days
  A serum createnine-based modification of the Acute Kidney Injury Network criteria:
  Stage 0: No change in SCr, Stage 1:↑SCr 0.3 mg/dL or ↑SCr 150- <200% from previous trough value, Stage 2: ↑ SCr 200- <300% from previous trough value, Stage 3: ↑ SCr ≥300% from previous trough value, SCr 2.5 mg/dL, or dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, El Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nour I, Elmaghraby R, Shehata R, El-Refaey A, Aldomiaty H, Mosbah A, Shouman B, Nasef N. Selective head cooling and acute kidney injury in neonates with hypoxic ischemic encephalopathy. J Neonatal Perinatal Med. 2020;13(1):21-30. doi: 10.3233/NPM-180200. PMID 31561395